CLINICAL TRIAL: NCT00840892
Title: Randomized Controlled Trial to Establish the (Cost-)Effectiveness of an Interdisciplinary Community-based COPD Management Program Relative to Usual Care.
Brief Title: (Cost-)Effectiveness Interdisciplinary Community-based COPD Management Program (INTERCOM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maxima Medical Center (Other); Erasmus Medical Center (Other); The Netherlands Asthma Foundation (Other); Stichting Astma Bestrijding, The Netherlands (Other); Nutricia Netherlands (Unknown); PICASSO: Partners in Care Solutions for COPD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERCOM_CCMO_P00.1631L; Neth Asthma Found., 3.4.01.63
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2009-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intercom (Experimental): INTERdisciplinary COMmunity-based COPD management (INTERCOM)
  Interventions: Other: INTERdisciplinary COMmunity-based COPD management (INTERCOM)
- Usual Care (No Intervention)

INTERVENTIONS:
Other: INTERdisciplinary COMmunity-based COPD management (INTERCOM) — The INTERCOM program consisted of exercise training, education, nutritional therapy and smoking cessation support offered by local physiotherapists and dieticians in the proximity of the patient's home and by respiratory nurses in the hospital. The program was divided in a 4-month intensive intervention phase, followed by a 20-month maintenance phase.
  Arms: Intercom

SUMMARY:
There is growing evidence that COPD is a multi-organ system disease. Besides impaired lung function, skeletal muscle weakness and weight loss are important determinants of impaired exercise performance, decreased quality of life and increased mortality. Based on earlier succesful intervention studies in pulmonary rehabilitation settings, Máxima Medical Centre developed an integrated, inter-disciplinary approach to the management of COPD including physical exercise, nutritional therapy, education, smoking cessation and psychological consultation. This COPD management program consists of a set of protocols that cover patient recruitment, diagnostic testing, treatment, follow-up and communication between professionals.

The exercise program and the nutitional therapy are carried out by local physiotherapists and dieticians working outside but in conjunction with the hospital. A program in such a setting could be substantially less expensive and certainly more easily accessible for many more patients than an inpatient or hospital-based outpatient rehabilitation program, as it is offered close to a patient's home. This study investigates the (cost-)effectiveness of the COPD management program compared to usual care in a randomized controlled trial.

Patients with moderate to severe COPD and a reduced exercise capacity during an incremental exercise test of less than 70% of predicted, are randomised to a treatment or a control group. The treatment group will participate in the COPD management program during the first 4 months after which they will be followed up for the remaining months. Both groups (n=100) are followed for 2 years and outcomes will be assessed at the beginning of the program, after 4, 12 and 24 months by disease-specific and generic measures of health status, body composition, skeletal muscle function and exercise capacity. A cost-effectiveness and cost-utility analysis with a two-year time horizon will be performed. The analysis is conducted from a societal perspectice, including the program costs and all COPD-related direct costs within and outside the healthcare sector ans costs of lost productivity.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD according to the recent GOLD guidelines
* Reduced exercise capacity during an incremental exercise test of less than 70% of predicted normal values

Exclusion Criteria:

* Lack of motivation to participate in the treatment program
* Other pathologic conditions unabling participation in the training program (e.g. coronary, orthopaedic, neurological or severe endocrine disorders)
* participation in other pulmonary rehabilitation projects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2002-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The two primary outcomes are disease-specific quality of life assessed with the St. George's Respiratory Questionnaire (SGRQ) and the total number of exacerbations

SECONDARY OUTCOMES:
dyspnea, quality of life, exercise performance measures, body composition measures and lung function

CONTACTS AND LOCATIONS:
Overall Officials: Annemie MWJ Schols, Prof PhD, Principal Investigator — Maastricht University Medical Centre
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - Maxima Medical Centre, Veldhoven/Eindhoven

REFERENCES:
- [Derived] van Wetering CR, Hoogendoorn M, Broekhuizen R, Geraerts-Keeris GJ, De Munck DR, Rutten-van Molken MP, Schols AM. Efficacy and costs of nutritional rehabilitation in muscle-wasted patients with chronic obstructive pulmonary disease in a community-based setting: a prespecified subgroup analysis of the INTERCOM trial. J Am Med Dir Assoc. 2010 Mar;11(3):179-87. doi: 10.1016/j.jamda.2009.12.083. Epub 2010 Feb 4. PMID 20188315
- [Derived] van Wetering CR, Hoogendoorn M, Mol SJ, Rutten-van Molken MP, Schols AM. Short- and long-term efficacy of a community-based COPD management programme in less advanced COPD: a randomised controlled trial. Thorax. 2010 Jan;65(1):7-13. doi: 10.1136/thx.2009.118620. Epub 2009 Aug 23. PMID 19703824
- [Derived] Hoogendoorn M, van Wetering CR, Schols AM, Rutten-van Molken MP. Is INTERdisciplinary COMmunity-based COPD management (INTERCOM) cost-effective? Eur Respir J. 2010 Jan;35(1):79-87. doi: 10.1183/09031936.00043309. Epub 2009 Jul 2. PMID 19574331